CLINICAL TRIAL: NCT03013400
Title: A Randomised, Parallel Group, Double Blind, Placebo Controlled, Add on Clinical Trial to Investigate Whether the Lithium Mimetic, Ebselen, Can Reduce Symptoms of Hypomania and Mania in Bipolar Patients
Brief Title: Ebselen as an add-on Treatment in Hypo/Mania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Stanley Medical Research Institute (Other); Sound Pharmaceuticals, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 172518; 2015-000323-86 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2017-01-06 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2017-11

CONDITIONS: Bipolar Disorder; Bipolar Disorder, Manic
MeSH Terms: conditions — Bipolar Disorder | interventions — ebselen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ebselen (Active Comparator): Three Ebselen capsules each containing 200mg taken orally twice a day for 3 weeks
  Interventions: Drug: Ebselen
- Placebo (Placebo Comparator): Three Placebo capsules each containing 200mg taken orally twice a day for 3 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ebselen — Ebselen is an opaque capsule containing 200 mg of ebselen is a selenium-based GPx mimic and IMPase inhibitor.
  Other Names: SPI-1005; PZ-51; Ebselene; Ebselenum; Ebseleno; Harmokisane
  Arms: Ebselen
Drug: Placebo oral capsule — Placebo is identical in appearance to the ebselen capsules
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
This study evaluates the effect of a 'lithium like' drug called ebselen (SP-1005) versus placebo as an 'add on' treatment to help stabilise hypo/manic symptoms in bipolar disorder. Half of the participants will receive ebselen and the other half placebo. The trial, will last a total of four weeks.

DETAILED DESCRIPTION:
Ebselen, a new drug for mania

Bipolar disorder, formerly known as manic depression, is a condition that affects mood, which can swing from one extreme to another.

Typically, there will be periods of:

* Depression - very low mood and energy levels
* Mania or hypomania (less severe) - very high mood and overactive energy levels

A drug called lithium, used to stabilise mood, is an important treatment for bipolar disorder but has a number of problematic side effects, is not well tolerated by patients and requires careful monitoring. To replace lithium with other, safer medicines would have clear advantages. The investigators are interested in an antioxidant medicine(substance that may prevent or delay cell damage) called ebselen which has been shown to work in a similar way as lithium and the investigators are investigating whether it might help improve recovery from manic episodes.

The present study aims to see whether ebselen, used as an 'add-on' treatment can help stabilise mood in patients experiencing high mood (hypo/mania). Sixty patients experiencing hypo/mania will be given in a randomised order (similar to tossing a coin) either ebselen or placebo (dummy) in addition to their usual medication for three weeks after which the add-on treatment will be stopped. A final follow up visit will take place one week after the study medication has been stopped. Participants can be in or outpatients and mood will be monitored with questionnaires and interviews. Activity will also be monitored with the use of an actiwatch (similar to a wrist watch) which will be worn continuously throughout the study. A single blood sample will be optional and occur after the first week of treatment to check plasma levels of ebselen and inflammatory markers. A positive outcome in this trial will be followed by longer term studies of ebselen in bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18-70 years
* Diagnosed with bipolar disorder, screened using the Structured Clinical Interview for DSM-5 (SCID) to meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for Manic or Hypomanic Episode.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow clinical care team (including General Practitioner (GP)) to be made aware of trial participation.
* The Clinical team treating the patient are in agreement.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Known significant renal or hepatic impairment.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Clinically significant illicit substance or alcohol misuse where dependence criteria are satisfied.
* Taking lithium.
* Previous randomisation to this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) | Change between groups, every week, up to 4 weeks
  Difference in the 11 item clinician-rated YMRS between groups.Total score 0-60.

SECONDARY OUTCOMES:
Change in Clinical Global Impressions Bipolar (CGI-BP) mania scale | Change between groups, every week, up to 4 weeks
  Improvement due to treatment between groups. Very much improved to very much worse.
Change in Altman Self Rating Mania Scale (ASRM) | Change between groups, 3 x weekly, up to 4 weeks
  Difference in the 5 item self-rated ASRM between groups.Total score 0-20.
Change in Hamilton Rating Scale for Depression (HAM-D) | Change between groups, every week, up to 4 weeks
  Difference in the 17 item Clinician-rated HAM-D between groups. Total score 0-52.
Change in Quick Inventory of Depressive Symptomology-Self Rating 16 (QIDS-SR-16) | Change between groups, 3 x weekly, up to 4 weeks
  Difference in the 16 item self-rated QIDS-SR-16 between groups. Total score 0-42.
Change in Actigraphy | Change in activity between groups, each 24 hours, up to 4 weeks
  To compare the effect of ebselen versus placebo on motor behaviour and the sleep-wake cycle
Change in Leeds Sleep Evaluation Questionnaire (LSEQ) | Change between groups, every week, up to 4 weeks
  Difference in the 4 self-rated sleep domains (10 visual analogue scales) between groups.
Levels of markers of inflammation in Plasma sample | Once at week 1 visit
  To compare the effect of ebselen, versus placebo, on markers of inflammation including C-Reactive Protein and antibodies to common infectious agents such as human herpesviruses and Toxoplasma gondii
Ebselen levels in Plasma sample | Once at week 1 visit
  To assess ebselen levels in plasma
Adverse Events reported | Every week, up to 4 weeks
  Self-rated Side Effects Questionnaire
Change in Concomitant medication recorded | Change between groups, every week, up to 4 weeks
  To assess the overall use of concomitant medication during the trial period
Compliance assessment | Change between groups, every week, up to 3 weeks
  capsule count and records checked

OTHER OUTCOMES:
Researcher and participant blinding questionnaire to determine treatment concealment | Once, at week 4
  Researcher and participant blinding questionnaire
Participant and Researcher Randomisation Guess Visual Analogue Scale (VAS) | Once, at week 4
  To assess whether researchers and participants could guess the assigned randomised arm
Public Participant Involvement (PPI) feedback questionnaire | Once, at week 4
  PPI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cowen, MBBS, MD, Principal Investigator — University of Oxford
Locations (1):
- Neurosciences Building, Dept. Psychiatry, Warneford Hospital, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Masaki C, Sharpley AL, Cooper CM, Godlewska BR, Singh N, Vasudevan SR, Harmer CJ, Churchill GC, Sharp T, Rogers RD, Cowen PJ. Effects of the potential lithium-mimetic, ebselen, on impulsivity and emotional processing. Psychopharmacology (Berl). 2016 Jul;233(14):2655-61. doi: 10.1007/s00213-016-4319-5. Epub 2016 Jun 2. PMID 27256357
- [Background] Masaki C, Sharpley AL, Godlewska BR, Berrington A, Hashimoto T, Singh N, Vasudevan SR, Emir UE, Churchill GC, Cowen PJ. Effects of the potential lithium-mimetic, ebselen, on brain neurochemistry: a magnetic resonance spectroscopy study at 7 tesla. Psychopharmacology (Berl). 2016 Mar;233(6):1097-104. doi: 10.1007/s00213-015-4189-2. Epub 2016 Jan 12. PMID 26758281
- [Background] Singh N, Sharpley AL, Emir UE, Masaki C, Herzallah MM, Gluck MA, Sharp T, Harmer CJ, Vasudevan SR, Cowen PJ, Churchill GC. Effect of the Putative Lithium Mimetic Ebselen on Brain Myo-Inositol, Sleep, and Emotional Processing in Humans. Neuropsychopharmacology. 2016 Jun;41(7):1768-78. doi: 10.1038/npp.2015.343. Epub 2015 Nov 23. PMID 26593266
- [Background] Singh N, Halliday AC, Thomas JM, Kuznetsova OV, Baldwin R, Woon EC, Aley PK, Antoniadou I, Sharp T, Vasudevan SR, Churchill GC. A safe lithium mimetic for bipolar disorder. Nat Commun. 2013;4:1332. doi: 10.1038/ncomms2320. PMID 23299882
- [Derived] Sharpley AL, Williams C, Holder AA, Godlewska BR, Singh N, Shanyinde M, MacDonald O, Cowen PJ. A phase 2a randomised, double-blind, placebo-controlled, parallel-group, add-on clinical trial of ebselen (SPI-1005) as a novel treatment for mania or hypomania. Psychopharmacology (Berl). 2020 Dec;237(12):3773-3782. doi: 10.1007/s00213-020-05654-1. Epub 2020 Sep 9. PMID 32909076
- [Derived] Garland M, Hryckowian AJ, Tholen M, Bender KO, Van Treuren WW, Loscher S, Sonnenburg JL, Bogyo M. The Clinical Drug Ebselen Attenuates Inflammation and Promotes Microbiome Recovery in Mice after Antibiotic Treatment for CDI. Cell Rep Med. 2020 Apr 21;1(1):100005. doi: 10.1016/j.xcrm.2020.100005. PMID 32483557